CLINICAL TRIAL: NCT01927861
Title: A 52-week, Multi-centre, Randomised, Double-blind, Parallel-group, no Treatment Controlled (Open-label) Trial Investigating the Efficacy and Safety of Two Doses of NN-220 in Short Stature With Noonan Syndrome
Brief Title: Investigating the Long-term Efficacy and Safety of Two Doses of NN-220 (Somatropin) in Short Stature Due to Noonan Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GHLIQUID-4020; U1111-1131-5892 (Other: WHO); JapicCTI-132336 (Registry Identifier: JAPIC)
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Results first posted 2019-10-14 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: Genetic Disorder; Noonan Syndrome
MeSH Terms: conditions — Genetic Diseases, Inborn; Noonan Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.033 mg/kg/day (Experimental)
  Interventions: Drug: somatropin
- 0.066 mg/kg/day (Experimental)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Administered subcutaneously (s.c., under the skin) in a daily regimen for at least 104 weeks. Subject will be offered to continue treatment for another 104 weeks.

SUMMARY:
This trial is conducted in Asia. The aim of the trial is to investigate the long-term efficacy and safety of two doses of NN-220 (somatropin) in short stature due to Noonan syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Japanese children with Noonan syndrome clinically diagnosed in one of the following ways: 1. Clinically diagnosed by at least two medical experts using van der Burgt score list, 2. Clinically diagnosed by one medical expert using van der Burgt score list and diagnosed by result of genetic testing for Noonan syndrome, 3. Clinically diagnosed by one medical expert using van der Burgt score list and diagnosed by the same medical expert based on the results of centralised evaluation of facial change using van der Burgt score list
* Height SDS (standard deviation score): -2 SDS or below (according to the Japanese reference data)
* Age: boys 3 to below 11 years, girls 3 to below 10 years
* Height records must be available within the period between 40 and 64 weeks prior to Visit 1 (screening)
* Prepubertal children (definition for girls breast and pubes of Tanner stage is I, and none of menses, and for boys testicular volume below 4 mL, and pubes and penis of Tanner stage is I)

Exclusion Criteria:

* Children with known or suspected hypersensitivity against human growth hormone (hGH) or related products (including any components of the trial products)
* Children with diabetic type diagnosed with the Japanese Diabetes Society Classification
* Children with history or presence of active malignancy
* Children who have received GH (growth hormone) treatment
* Children who have received systemic administration of the following medications within two years prior to Visit 1 (screening): Thyroid hormone (except replacement therapy), antithyroid hormone, androgen, oestrogen, progesterone, anabolic steroid, adrenocortical steroid treatment period for at least 13 weeks), derivative of gonadotropin releasing hormone and somatomedin C (IGF-I)

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2013-08-19 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (19):
- Japan (19):
  - Novo Nordisk Investigational Site, Asahikawa, Hokkaido
  - Novo Nordisk Investigational Site, Fukuoka
  - Novo Nordisk Investigational Site, Iruma-gun, Saitama
  - Novo Nordisk Investigational Site, Kanagawa
  - Novo Nordisk Investigational Site, Kyoto
  - Novo Nordisk Investigational Site, Maebashi-shi, Gunma
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Nagoya, Aichi
  - Novo Nordisk Investigational Site, Niigata-shi, Niigata
  - Novo Nordisk Investigational Site, Osaka
  - Novo Nordisk Investigational Site, Ōita
  - Novo Nordisk Investigational Site, Saitama-city, Saitama
  - Novo Nordisk Investigational Site, Saitama-shi, Saitama
  - Novo Nordisk Investigational Site, Sapporo, Hokkaido
  - Novo Nordisk Investigational Site, Sendai-shi, Miyagi
  - Novo Nordisk Investigational Site, Shizuoka
  - Novo Nordisk Investigational Site, Tochigi
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Zentsuji, Kagawa

REFERENCES:
- [Result] Horikawa R, Ogata T, Matsubara Y, Yokoya S, Ogawa Y, Nishijima K, Endo T, Ozono K. Long-term efficacy and safety of two doses of Norditropin(R) (somatropin) in Noonan syndrome: a 4-year randomized, double-blind, multicenter trial in Japanese patients. Endocr J. 2020 Aug 28;67(8):803-818. doi: 10.1507/endocrj.EJ19-0371. Epub 2020 May 9. PMID 32269181
- [Result] Ozono K, Ogata T, Horikawa R, Matsubara Y, Ogawa Y, Nishijima K, Yokoya S. Efficacy and safety of two doses of Norditropin(R) (somatropin) in short stature due to Noonan syndrome: a 2-year randomized, double-blind, multicenter trial in Japanese patients. Endocr J. 2018 Feb 26;65(2):159-174. doi: 10.1507/endocrj.EJ17-0313. Epub 2017 Nov 7. PMID 29109363
- [Derived] Muroya K, Kawai M, Yamagishi H, Endo T, Pietropoli A, Ferran JM, Horikawa R. Long-term effectiveness and safety of daily growth hormone therapy in Japanese children with Noonan syndrome: a post-marketing surveillance study. Endocr J. 2025 Nov 22. doi: 10.1507/endocrj.EJ25-0116. Online ahead of print. PMID 41285480
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 26 sites in Japan.
Pre-assignment Details: Participants were assigned to treatment for 104 weeks in the pivotal phase and for further 104 weeks in the extension phase and were offered to continue treatment in the extended treatment phase for 26 weeks.
Groups:
- NN-220 0.033 mg/kg/Day: Participants received subcutaneous (s.c.) injection of NN-220, 0.033 milligrams per kilogram per day (mg/kg/day) once daily for 234 weeks (104 weeks of pivotal phase + 104 weeks of extension phase + 26 weeks extended treatment phase).
- NN-220 0.066 mg/kg/Day: Participants received s.c. injection of NN-220, 0.066 mg/kg/day once daily for 234 weeks (104 weeks of pivotal phase + 104 weeks of extension phase + 26 weeks extended treatment phase).
Period: Pivotal Phase (104 Weeks)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Started | 25 | 26
Completed | 25 | 26
Not Completed | 0 | 0
Period: Extension Phase (104 Weeks)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Started | 25 | 26
Completed | 25 | 23
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Unclassified | 0 | 1
Period: Extended Treatment Phase (26 Weeks)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Started | 15 (15 participants agreed to continue the treatment for 26 weeks in the extended treatment phase.) | 14 (14 participants agreed to continue the treatment for 26 weeks in the extended treatment phase.)
Completed | 15 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) which included all randomised participants.
Groups:
- NN-220 0.033 mg/kg/Day: Participants received s.c. injection of NN-220, 0.033 mg/kg/day once daily for 234 weeks (104 weeks of pivotal phase + 104 weeks of extension phase + 26 weeks extended treatment phase).
- Total: Total of all reporting groups
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.57 (2.42) | 6.06 (2.25) | 6.31 (2.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 14 | 18 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 25 | 26 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height standard deviation score (SDS) (Japanese national reference data) [Mean (Standard Deviation); unit: Standard deviation score] — Height SDS was calculated using the formula: SDS = (height - mean)/SD, where height was the height variable measured, mean and standard deviation (SD) of height by sex and age for the reference population. The scores were centered around zero. Positive SDS indicated greater height and negative SDS indicated lesser height than the mean of the reference population.
  Standard deviation score | -3.24 (0.76) | -3.25 (0.71) | -3.24 (0.73)

OUTCOME MEASURES:

1. Primary Outcome: Change in Height SDS (Japanese National Reference Data)
Description: Height SDS was calculated using the formula: SDS = (height - mean)/SD, where height was the height variable measured, mean and SD of height by sex and age for the reference population. The scores were centered around zero. Positive SDS indicated greater height and negative SDS indicated lesser height than the mean of the reference population. The change from baseline (week 0) in the height SDS after 104 weeks of treatment was analysed using an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline height SDS as a covariate. Positive value in change from baseline indicated that SDS was better than baseline SDS. Missing values were imputed using the last observation carried forward (LOCF) method.
Time Frame: Baseline, week 104
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: Standard deviation score
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Standard deviation score | 0.84 (0.09) | 1.47 (0.09)
Statistical Analysis 1: Comparison: NN-220 0.033 mg/kg/Day vs NN-220 0.066 mg/kg/Day; The change from baseline (week 0) in the height SDS after 104 weeks of treatment was analysed using an ANCOVA model with treatment as a fixed effect and baseline height SDS as a covariate; Test type: Other; p < 0.0001, ANCOVA; Treatment difference = 0.63, 95% CI 2-sided [0.38 to 0.88]

2. Secondary Outcome: Height Velocity SDS
Description: Height velocity is change in height per year. The height velocity was calculated as the difference between current height (week 52) and height at baseline (week 0) divided by time between those measurement time points and multiplied by 365 days. Height velocity SDS was calculated using the formula: SDS = (height velocity - mean)/SD, where height velocity was the height velocity variable measured, mean and SD of height velocity by sex and age for the reference population. The scores were centered around zero. Positive SDS indicated greater height velocity and negative SDS indicated lesser height velocity than the mean of the reference population.
Time Frame: Baseline to week 52
Population: FAS.
Measure: Mean (Standard Deviation); unit: Standard deviation score
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Standard deviation score | 2.80 (1.13) | 5.01 (1.92)

3. Secondary Outcome: Height Velocity SDS
Description: Height velocity is change in height per year. The height velocity was calculated as the difference between current height (week 104) and height at week 52 divided by time between those measurement time points and multiplied by 365 days. Height velocity SDS was calculated using the formula: SDS = (height velocity - mean)/SD, where height velocity was the height velocity variable measured, mean and SD of height velocity by sex and age for the reference population. The scores were centered around zero. Positive SDS indicated greater height velocity and negative SDS indicated lesser height velocity than the mean of the reference population.
Time Frame: Week 52 to week 104
Population: FAS.
Measure: Mean (Standard Deviation); unit: Standard deviation score
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Standard deviation score | 0.58 (1.59) | 2.65 (1.76)

4. Secondary Outcome: Height Velocity
Description: Height velocity is change in height per year. The height velocity was calculated as the difference between current height (week 52) and height at baseline (week 0) divided by time between those measurement time points and multiplied by 365 days.
Time Frame: Baseline to week 52
Population: FAS.
Measure: Mean (Standard Deviation); unit: Centimeters per year (cm/year)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Centimeters per year (cm/year) | 7.88 (0.87) | 9.90 (1.49)

5. Secondary Outcome: Height Velocity
Description: Height velocity is change in height per year. The height velocity was calculated as the difference between current height (week 104) and height at week 52 divided by time between those measurement time points and multiplied by 365 days.
Time Frame: Week 52 to week 104
Population: FAS.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
cm/year | 6.20 (0.95) | 7.99 (1.20)

6. Secondary Outcome: Incidence of Treatment Emergent Adverse Events
Description: A treatment emergent adverse event (TEAE; for the pivotal phase) was defined as an event that had onset date on or after the date of visit 2 (week 0; start of treatment) and no later than the date of visit 12 (104 weeks; end of pivotal phase). For withdrawal participants (if any), an adverse event with onset date no later than 7 days after the last day of NN-220 treatment was included.
Time Frame: During 104 weeks of treatment
Population: Safety analysis set (SAS) which included all participants who received at least one dose of trial product (NN-220, 0.033 mg/kg/day or NN-220, 0.066 mg/kg/day).
Measure: Number; unit: Events
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Events | 265 | 306

7. Secondary Outcome: Change in IGF-I (Insulin-like Growth Factor-I)
Description: Change from baseline (within 4 weeks prior to week 0) in IGF-I was evaluated after 104 weeks of treatment. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 104
Population: SAS.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Nanograms per milliliter (ng/mL) | 90.4 (65.5) | 159.1 (88.0)

8. Secondary Outcome: Change in HbA1c (Glycosylated Haemoglobin)
Description: Change from baseline (within 4 weeks prior to week 0) in HbA1c was evaluated after 104 weeks of treatment.
Time Frame: Baseline, week 104
Population: SAS.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Percentage of HbA1c | 0.14 (0.18) | 0.13 (0.20)

9. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Erythrocytes)
Description: Change from baseline (within 4 weeks prior to week 0) in haematological parameter - erythrocytes. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 104
Population: SAS.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (10^12 cells/L)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
10^12 cells per liter (10^12 cells/L) | 0.106 (0.300) | 0.165 (0.234)

10. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Leukocytes and Thrombocytes)
Description: Change from baseline (within 4 weeks prior to week 0) in haematological parameter - leukocytes and thrombocytes. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 104
Population: SAS. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (10^9 cells/L)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
10^9 cells per liter (10^9 cells/L)
  Leukocytes | -0.69 (2.28) | -1.01 (1.77)
  Thrombocytes: number analyzed (Participants) | 24 | 26
  Thrombocytes | -6.9 (60.2) | -29.0 (63.2)

11. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Haemoglobin)
Description: Change from baseline (within 4 weeks prior to week 0) in haematological parameter - haemoglobin. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 104
Population: SAS.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Millimoles per liter (mmol/L) | 0.26 (0.46) | 0.32 (0.55)

12. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Haematocrit)
Description: Change from baseline (within 4 weeks prior to week 0) in haematological parameter - haematocrit. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 104
Population: SAS.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Percentage of red blood cells | 0.85 (2.11) | 0.94 (1.93)

13. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Neutrophils)
Description: Change from baseline (within 4 weeks prior to week 0) in haematological parameter - neutrophils. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 104
Population: SAS.
Measure: Mean (Standard Deviation); unit: Percentage of neutrophils
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Percentage of neutrophils | -4.28 (11.44) | 4.50 (9.01)

14. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Lymphocytes)
Description: Change from baseline (within 4 weeks prior to week 0) in haematological parameter - lymphocytes. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 104
Population: SAS.
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Percentage of lymphocytes | 2.80 (9.07) | -4.73 (8.73)

15. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Monocytes)
Description: Change from baseline (within 4 weeks prior to week 0) in haematological parameter - monocytes. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 104
Population: SAS.
Measure: Mean (Standard Deviation); unit: Percentage of monocytes
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Percentage of monocytes | 0.38 (1.41) | 0.39 (1.35)

16. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Eosinophils)
Description: Change from baseline (within 4 weeks prior to week 0) in haematological parameter - eosinophils. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 104
Population: SAS.
Measure: Mean (Standard Deviation); unit: Percentage of eosinophils
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Percentage of eosinophils | 0.99 (2.95) | -0.05 (1.33)

17. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Basophils)
Description: Change from baseline (within 4 weeks prior to week 0) in haematological parameter - basophils. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 104
Population: SAS.
Measure: Mean (Standard Deviation); unit: Percentage of basophils
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Percentage of basophils | 0.10 (0.36) | -0.07 (0.27)

18. Secondary Outcome: Change in Clinical Laboratory Tests (Lipids: Total Cholesterol, LDL Cholesterol and HDL Cholesterol)
Description: Change from baseline (within 4 weeks prior to week 0) in lipids: total cholesterol, LDL (low-density lipoprotein) cholesterol and HDL (high-density lipoprotein) cholesterol. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 104
Population: SAS.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
mmol/L
  Total cholesterol | 0.073 (0.655) | -0.110 (0.371)
  LDL cholesterol | 0.040 (0.521) | -0.120 (0.323)
  HDL cholesterol | -0.020 (0.212) | -0.034 (0.210)

19. Secondary Outcome: Change in Clinical Laboratory Tests (Biochemistry: AST, ALT, r-GTP and Alkaline Phosphatase)
Description: Change from baseline (within 4 weeks prior to week 0) in biochemical parameters - aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyl transpeptidase (r-GTP) and alkaline phosphatase. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 104
Population: SAS. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Units per liter (U/L)
  AST: number analyzed (Participants) | 24 | 26
  AST | -3.6 (2.9) | -6.0 (4.3)
  ALT | -1.04 (3.10) | -1.73 (4.20)
  r-GTP | 0.4 (1.6) | -3.7 (19.4)
  Alkaline phosphatase: number analyzed (Participants) | 24 | 26
  Alkaline phosphatase | 73.8 (76.3) | 124.3 (124.0)

20. Secondary Outcome: Change in Clinical Laboratory Tests (Biochemistry: Total Protein)
Description: Change from baseline (within 4 weeks prior to week 0) in biochemical parameter - total protein. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 104
Population: SAS. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Grams per deciliter (g/dL)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Grams per deciliter (g/dL) | 0.02 (0.38) | -0.05 (0.27)

21. Secondary Outcome: Change in Clinical Laboratory Tests (Biochemistry: Blood Urea Nitrogen, Sodium, Potassium, Chloride, Total Calcium and Phosphorus)
Description: Change from baseline (within 4 weeks prior to week 0) in biochemical parameters - blood urea nitrogen, sodium, potassium, chloride, total calcium and phosphorus. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 104
Population: SAS. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
mmol/L
  Blood urea nitrogen | -0.17 (0.38) | -0.21 (0.44)
  Sodium | -0.3 (2.4) | -0.2 (2.6)
  Potassium: number analyzed (Participants) | 24 | 26
  Potassium | -0.03 (0.32) | -0.15 (0.41)
  Chloride | -0.8 (2.3) | -1.3 (1.9)
  Total calcium: number analyzed (Participants) | 24 | 26
  Total calcium | 0.00 (0.08) | 0.01 (0.07)
  Phosphorus: number analyzed (Participants) | 24 | 26
  Phosphorus | 0.124 (0.125) | 0.129 (0.141)

22. Secondary Outcome: Change in Clinical Laboratory Tests (Biochemistry: Creatinine)
Description: Change from baseline (within 4 weeks prior to week 0) in biochemical parameter - creatinine. Missing values were imputed using the LOCF method.
Time Frame: Baseline, Week 104
Population: SAS.
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Micromoles per liter (umol/L) | 1.8 (3.5) | 2.5 (3.4)

23. Secondary Outcome: Change in Glucose Tolerance (AUC of Glucose) Based on the OGTT
Description: AUC (area under the curve) of glucose was calculated by the trapezoidal method. Change from baseline (within 4 weeks prior to week 0) in glucose tolerance (AUC of glucose: 30, 60, 90 and 120 min after oral glucose load) at week 104 was evaluated based on the oral glucose tolerance test (OGTT). Change from baseline results are presented as 'ratio to baseline'.
Time Frame: Baseline, week 104
Population: SAS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Ratio of AUC | 0.98 (12.19) | 1.04 (17.75)

24. Secondary Outcome: Change in Glucose Tolerance (AUC of Insulin) Based on the OGTT
Description: AUC of insulin was calculated by the trapezoidal method. Change from baseline (within 4 weeks prior to week 0) in glucose tolerance (AUC of insulin: 30, 60, 90 and 120 min after oral glucose load) at week 104 was evaluated based on the OGTT. Change from baseline results are presented as 'ratio to baseline'.
Time Frame: Baseline, week 104
Population: SAS. Number analyzed = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Ratio of AUC | 1.25 (45.08) | 1.72 (85.78)

25. Secondary Outcome: Change in Bone Age
Description: X-ray picture of carpal bones of left hand was taken for bone age determination. Centralised evaluation of bone age was done by the radius, ulna and short bones (RUS) score method of Tanner-Whitehouse II (TW2). Change from baseline (week 0) in bone age.
Time Frame: Baseline, week 104
Population: SAS.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Years | 2.07 (0.80) | 2.63 (0.94)

26. Secondary Outcome: Change in Bone Age/Chronological Age
Description: X-ray picture of carpal bones of left hand was taken for bone age determination. Centralised evaluation of bone age was done by the RUS score method of Tanner-Whitehouse II (TW2). Change from baseline (week 0) in bone age/chronological age.
Time Frame: Baseline, week 104
Population: SAS.
Measure: Mean (Standard Deviation); unit: Ratio (bone age/chronological age)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Ratio (bone age/chronological age) | 0.047 (0.127) | 0.133 (0.127)

27. Secondary Outcome: Yearly Change in Bone Age/Change in Chronological Age
Description: X-ray picture of carpal bones of left hand was taken for bone age determination. Centralised evaluation of bone age was done by the RUS score method of Tanner-Whitehouse II (TW2). Yearly change from baseline (week 0) in bone age/change in chronological age was presented.
Time Frame: Baseline, week 52
Population: SAS.
Measure: Mean (Standard Deviation); unit: Ratio (bone age/chronological age)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Ratio (bone age/chronological age) | 0.93 (0.66) | 1.28 (0.70)

28. Secondary Outcome: Yearly Change in Bone Age/Change in Chronological Age
Description: X-ray picture of carpal bones of left hand was taken for bone age determination. Centralised evaluation of bone age was done by the RUS score method of Tanner-Whitehouse II (TW2). Yearly change from week 52 in bone age/change in chronological age was presented.
Time Frame: Week 52, week 104
Population: SAS.
Measure: Mean (Standard Deviation); unit: Ratio (bone age/chronological age)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Ratio (bone age/chronological age) | 1.15 (0.57) | 1.38 (0.91)

29. Secondary Outcome: Change in Vital Signs (Diastolic Blood Pressure and Systolic Blood Pressure)
Description: Systolic and diastolic blood pressure were measured after a 5-minute rest in sitting position. Change from baseline (week 0) in systolic blood pressure and diastolic blood pressure.
Time Frame: Baseline, week 104
Population: SAS. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Millimeters of mercury (mmHg)
  Diastolic blood pressure: number analyzed (Participants) | 25 | 25
  Diastolic blood pressure | 2.3 (13.2) | 6.3 (15.8)
  Systolic blood pressure: number analyzed (Participants) | 25 | 25
  Systolic blood pressure | 5.5 (11.9) | 4.1 (12.1)

30. Secondary Outcome: Change in Vital Signs (Pulse)
Description: Pulse was measured after a 5-minute rest in sitting position. Change from baseline (week 0) in pulse.
Time Frame: Baseline, week 104
Population: SAS. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Beats per minute (beats/min)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Beats per minute (beats/min) | -9.5 (15.7) | 1.8 (21.9)

31. Secondary Outcome: Change in Urinalysis (Protein, Glucose and Occult Blood)
Description: The urinalysis was the measurements of protein, glucose, and occult blood at baseline (within 4 weeks prior to week 0) and week 104 and categorised as negative, trace, 1+, 2+ and 3+. Missing values were imputed using the LOCF method. Number of participants in each category at baseline and week 104 are presented.
Time Frame: Baseline, week 104
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Participants
  Protein: Negative (Baseline) | 23 | 22
  Protein: Trace (Baseline) | 2 | 4
  Protein: 1+ (Baseline) | 0 | 0
  Protein: 2+ (Baseline) | 0 | 0
  Protein: 3+ (Baseline) | 0 | 0
  Protein: Negative (Week 104) | 18 | 16
  Protein: Trace (Week 104) | 7 | 8
  Protein: 1+ (Week 104) | 0 | 2
  Protein: 2+ (Week 104) | 0 | 0
  Protein: 3+ (Week 104) | 0 | 0
  Glucose: Negative (Baseline) | 25 | 26
  Glucose: Trace (Baseline) | 0 | 0
  Glucose: 1+ (Baseline) | 0 | 0
  Glucose: 2+ (Baseline) | 0 | 0
  Glucose: 3+ (Baseline) | 0 | 0
  Glucose: Negative (Week 104) | 25 | 26
  Glucose: Trace (Week 104) | 0 | 0
  Glucose: 1+ (Week 104) | 0 | 0
  Glucose: 2+ (Week 104) | 0 | 0
  Glucose: 3+ (Week 104) | 0 | 0
  Occult blood: Negative (Baseline) | 24 | 25
  Occult blood: Trace (Baseline) | 1 | 1
  Occult blood: 1+ (Baseline) | 0 | 0
  Occult blood: 2+ (Baseline) | 0 | 0
  Occult blood: 3+ (Baseline) | 0 | 0
  Occult blood: Negative (Week 104) | 25 | 20
  Occult blood: Trace (Week 104) | 0 | 5
  Occult blood: 1+ (Week 104) | 0 | 0
  Occult blood: 2+ (Week 104) | 0 | 1
  Occult blood: 3+ (Week 104) | 0 | 0

32. Secondary Outcome: Change in Blood Coagulation Test (Prothrombin Time and APTT)
Description: Change from baseline (within 4 weeks prior to week 0) in blood coagulation test parameters: Prothrombin time and APTT (activated partial thromboplastin time). Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 104
Population: SAS.
Measure: Median (Full Range); unit: Second (sec)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Second (sec)
  Prothrombin time | 0.50 [-1.8 to 2.3] | 0.80 [-0.6 to 2.3]
  APTT | 0.60 [-4.0 to 4.7] | 0.25 [-9.1 to 5.6]

33. Secondary Outcome: Change in ECG
Description: The ECG was recorded after a 3-minute rest in supine position at baseline (within 4 weeks prior to week 0) and week 104 and categorised as normal, abnormal NCS (not clinically significant) or abnormal CS (clinically significant). Number of participants in each ECG category at baseline and week 104 are presented. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 104
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Participants
  Normal (Baseline) | 15 | 14
  Abnormal NCS (Baseline) | 10 | 12
  Abnormal CS (Baseline) | 0 | 0
  Normal (Week 104) | 16 | 13
  Abnormal NCS (Week 104) | 9 | 13
  Abnormal CS (Week 104) | 0 | 0

34. Secondary Outcome: Change in Height SDS (Japanese National Reference Data)
Description: Height SDS was calculated using the formula: SDS = (height - mean)/SD, where height was the height variable measured, mean and SD of height by sex and age for the reference population. The scores were centered around zero. Positive SDS indicated greater height and negative SDS indicated lesser height than the mean of the reference population. The change from baseline (week 0) in the height SDS after 208 weeks of treatment was analysed. Positive value in change from baseline indicated that SDS was better than baseline SDS. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 208
Population: FAS.
Measure: Mean (Standard Deviation); unit: Standard deviation score
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Standard deviation score | 0.85 (0.60) | 1.84 (0.70)

35. Secondary Outcome: Change in Height SDS (Noonan Syndrome Reference Data in Japanese)
Description: Height SDS was calculated using the formula: Z=[(value/M)^L-1]/(S*L); where L, M and S are skewness (L), median (M) and coefficient of variation (S) of Japanese Noonan syndrome' height provided for each sex and age. For each participant, a standard deviation score Z (SDS) was calculated based on age and sex referring to the values L, M and S. The scores were centered around zero. Positive SDS indicated greater height and negative SDS indicated lesser height than the mean of the reference population. The change from baseline (week 0) in the height SDS after 208 weeks of treatment was analysed. Positive value in change from baseline indicated that SDS was better than baseline SDS. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 208
Population: FAS.
Measure: Mean (Standard Deviation); unit: Standard deviation score
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Standard deviation score | 0.96 (0.47) | 1.92 (0.60)

36. Secondary Outcome: Height Velocity
Description: Height velocity is change in height per year. The height velocity was calculated as the difference between current height (week 156) and height at week 104 divided by time between those measurement time points and multiplied by 365 days. Missing values were imputed using the LOCF method.
Time Frame: Week 104 to week 156
Population: FAS.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
cm/year | 5.77 (1.26) | 7.01 (1.12)

37. Secondary Outcome: Height Velocity
Description: Height velocity is change in height per year. The height velocity was calculated as the difference between current height (week 208) and height at week 156 divided by time between those measurement time points and multiplied by 365 days. Missing values were imputed using the LOCF method.
Time Frame: Week 156 to week 208
Population: FAS.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
cm/year | 5.64 (1.23) | 6.11 (1.28)

38. Secondary Outcome: Height Velocity SDS
Description: Height velocity is change in height per year. The height velocity was calculated as the difference between current height (week 156) and height at week 104 divided by time between those measurement time points and multiplied by 365 days. Height velocity SDS was calculated using the formula: SDS = (height velocity - mean)/SD, where height velocity was the height velocity variable measured, mean and SD of height velocity by sex and age for the reference population. The scores were centered around zero. Positive SDS indicated greater height velocity and negative SDS indicated lesser height velocity than the mean of the reference population.
Time Frame: Week 104 to week 156
Population: FAS.
Measure: Mean (Standard Deviation); unit: Standard deviation score
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Standard deviation score | -0.39 (1.61) | 1.44 (1.25)

39. Secondary Outcome: Height Velocity SDS
Description: Height velocity is change in height per year. The height velocity was calculated as the difference between current height (week 208) and height at week 156 divided by time between those measurement time points and multiplied by 365 days. Height velocity SDS was calculated using the formula: SDS = (height velocity - mean)/SD, where height velocity was the height velocity variable measured, mean and SD of height velocity by sex and age for the reference population. The scores were centered around zero. Positive SDS indicated greater height velocity and negative SDS indicated lesser height velocity than the mean of the reference population.
Time Frame: Week 156 to week 208
Population: FAS.
Measure: Mean (Standard Deviation); unit: Standard deviation score
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Standard deviation score | -0.73 (1.52) | 0.92 (1.69)

40. Secondary Outcome: Incidence of Treatment Emergent AEs
Description: A treatment emergent AE (TEAE) was defined as an event that had onset date on or after the date of visit 2 (week 0; start of treatment) and no later than 7 days after the last day of NN-220 treatment.
Time Frame: Week 0 to week 234 (208 weeks treatment period + 26 weeks extended treatment period) + 7 days (follow-up period)
Population: SAS.
Measure: Number; unit: Events
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Events | 507 | 539

41. Secondary Outcome: Change in IGF-I
Description: Change from baseline (within 4 weeks prior to week 0) in IGF-I was evaluated after 208 weeks of treatment. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 208
Population: SAS.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
ng/mL | 133.5 (97.6) | 217.2 (91.1)

42. Secondary Outcome: Change in HbA1c
Description: Change from baseline (within 4 weeks prior to week 0) in HbA1c was evaluated after 208 weeks of treatment.
Time Frame: Baseline, week 208
Population: SAS. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Percentage of HbA1c | 0.19 (0.13) | 0.20 (0.21)

43. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Erythrocytes)
Description: as for outcome 9
Time Frame: Baseline, week 208
Population: SAS.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
10^12 cells/L | 0.121 (0.328) | 0.095 (0.204)

44. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Leukocytes and Thrombocytes)
Description: as for outcome 10
Time Frame: Baseline, Week 208
Population: SAS. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
10^9 cells/L
  Leukocytes | -1.50 (2.22) | -1.50 (1.57)
  Thrombocytes: number analyzed (Participants) | 24 | 26
  Thrombocytes | -27.5 (55.5) | -56.6 (58.5)

45. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Haemoglobin)
Description: as for outcome 11
Time Frame: Baseline, week 208
Population: SAS.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
mmol/L | 0.46 (0.58) | 0.46 (0.35)

46. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Haematocrit)
Description: as for outcome 12
Time Frame: Baseline, week 208
Population: SAS.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Percentage of red blood cells | 1.24 (2.45) | 1.26 (1.63)

47. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Neutrophils)
Description: as for outcome 13
Time Frame: Baseline, week 208
Population: SAS.
Measure: Mean (Standard Deviation); unit: Percentage of neutrophils
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Percentage of neutrophils | -1.23 (10.80) | 4.88 (9.41)

48. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Lymphocytes)
Description: as for outcome 14
Time Frame: Baseline, week 208
Population: SAS.
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Percentage of lymphocytes | -0.14 (8.88) | -5.70 (8.86)

49. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Monocytes)
Description: as for outcome 15
Time Frame: Baseline, week 208
Population: SAS.
Measure: Mean (Standard Deviation); unit: Percentage of monocytes
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Percentage of monocytes | 0.08 (1.21) | 0.56 (1.18)

50. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Eosinophils)
Description: as for outcome 16
Time Frame: Baseline, week 208
Population: SAS.
Measure: Mean (Standard Deviation); unit: Percentage of eosinophils
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Percentage of eosinophils | 1.30 (3.57) | 0.42 (1.44)

51. Secondary Outcome: Change in Clinical Laboratory Tests (Haematology: Basophils)
Description: as for outcome 17
Time Frame: Baseline, week 208
Population: SAS.
Measure: Mean (Standard Deviation); unit: Percentage of basophils
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Percentage of basophils | -0.01 (0.26) | -0.12 (0.26)

52. Secondary Outcome: Change in Clinical Laboratory Tests (Lipids: Total Cholesterol, LDL Cholesterol and HDL Cholesterol)
Description: Change from baseline (within 4 weeks prior to week 0) in lipids: total cholesterol, LDL cholesterol and HDL cholesterol. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 208
Population: SAS.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
mmol/L
  Total cholesterol | 0.031 (0.639) | -0.110 (0.609)
  LDL cholesterol | -0.005 (0.550) | -0.173 (0.523)
  HDL cholesterol | 0.036 (0.275) | 0.056 (0.173)

53. Secondary Outcome: Change in Clinical Laboratory Tests (Biochemistry: AST, ALT, r-GTP and Alkaline Phosphatase)
Description: Change from baseline (within 4 weeks prior to week 0) in biochemical parameters - AST, ALT, r-GTP and alkaline phosphatase. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 208
Population: SAS. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
U/L
  AST: number analyzed (Participants) | 24 | 26
  AST | -5.4 (2.4) | -7.4 (5.2)
  ALT | -1.28 (2.65) | -1.81 (4.42)
  r-GTP | 1.0 (1.6) | -3.5 (22.8)
  Alkaline phosphatase: number analyzed (Participants) | 24 | 26
  Alkaline phosphatase | 113.9 (126.4) | 84.8 (140.9)

54. Secondary Outcome: Change in Clinical Laboratory Tests (Biochemistry: Total Protein)
Description: as for outcome 20
Time Frame: Baseline, week 208
Population: SAS. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
g/dL | 0.02 (0.33) | 0.05 (0.37)

55. Secondary Outcome: Change in Clinical Laboratory Tests (Biochemistry: Blood Urea Nitrogen, Sodium, Potassium, Chloride, Total Calcium and Phosphorus)
Description: as for outcome 21
Time Frame: Baseline, week 208
Population: SAS. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
mmol/L
  Blood urea nitrogen | -0.10 (0.52) | -0.15 (0.53)
  Sodium | 0.9 (2.1) | 1.4 (2.5)
  Potassium: number analyzed (Participants) | 24 | 26
  Potassium | -0.13 (0.28) | -0.09 (0.38)
  Chloride | -0.3 (2.2) | -0.2 (2.2)
  Total calcium: number analyzed (Participants) | 24 | 26
  Total calcium | -0.02 (0.07) | -0.00 (0.08)
  Phosphorus: number analyzed (Participants) | 24 | 26
  Phosphorus | 0.036 (0.111) | 0.111 (0.103)

56. Secondary Outcome: Change in Clinical Laboratory Tests (Biochemistry: Creatinine)
Description: Change from baseline (within 4 weeks prior to week 0) in biochemical parameters - creatinine. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 208
Population: SAS.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
umol/L | 5.5 (4.4) | 6.7 (4.1)

57. Secondary Outcome: Change in Glucose Tolerance (AUC of Glucose) Based on the OGTT
Description: AUC of glucose was calculated by the trapezoidal method. Change from baseline (within 4 weeks prior to week 0) in glucose tolerance (AUC of glucose: 30, 60, 90 and 120 min after oral glucose load) at week 208 was evaluated based on the OGTT. Change from baseline results are presented as 'ratio to baseline'.
Time Frame: Baseline, week 208
Population: SAS. Number analyzed = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Ratio of AUC | 1.03 (12.34) | 1.10 (14.55)

58. Secondary Outcome: Change in Glucose Tolerance (AUC of Insulin) Based on the OGTT
Description: AUC of insulin was calculated by the trapezoidal method. Change from baseline (within 4 weeks prior to week 0) in glucose tolerance (AUC of insulin: 30, 60, 90 and 120 min after oral glucose load) at week 208 was evaluated based on the OGTT. Change from baseline results are presented as 'ratio to baseline'.
Time Frame: Baseline, week 208
Population: SAS. Number analyzed = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Ratio of AUC | 1.52 (49.97) | 2.38 (47.04)

59. Secondary Outcome: Change in Bone Age
Description: X-ray picture of carpal bones of left hand was taken for bone age determination. Centralised evaluation of bone age was done by the RUS score method of Tanner-Whitehouse II (TW2). Change from baseline (week 0) in bone age.
Time Frame: Baseline, week 208
Population: SAS. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Years | 3.89 (1.35) | 4.68 (1.11)

60. Secondary Outcome: Change in Bone Age/Chronological Age
Description: as for outcome 26
Time Frame: Baseline, week 208
Population: SAS. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Ratio (bone age/chronological age)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Ratio (bone age/chronological age) | 0.049 (0.159) | 0.149 (0.151)

61. Secondary Outcome: Yearly Change in Bone Age/Change in Chronological Age
Description: X-ray picture of carpal bones of left hand was taken for bone age determination. Centralised evaluation of bone age was done by the RUS score method of Tanner-Whitehouse II (TW2). Yearly change from week 104 in bone age/change in chronological age was presented.
Time Frame: Week 104, week 156
Population: SAS. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Ratio (bone age/chronological age)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Ratio (bone age/chronological age) | 0.94 (0.70) | 0.97 (0.56)

62. Secondary Outcome: Yearly Change in Bone Age/Change in Chronological Age
Description: X-ray picture of carpal bones of left hand was taken for bone age determination. Centralised evaluation of bone age was done by the RUS score method of Tanner-Whitehouse II (TW2). Yearly change from week 156 in bone age/change in chronological age was presented.
Time Frame: Week 156, week 208
Population: SAS. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Ratio (bone age/chronological age)
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Ratio (bone age/chronological age) | 0.87 (0.55) | 1.05 (0.51)

63. Secondary Outcome: Change in Vital Signs (Diastolic Blood Pressure and Systolic Blood Pressure)
Description: Systolic and diastolic blood pressure were measured after a 5-minute rest in sitting position. Change from baseline (week 0) in systolic blood pressure and diastolic blood pressure. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 208
Population: SAS. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
mmHg
  Diastolic blood pressure: number analyzed (Participants) | 25 | 25
  Diastolic blood pressure | 5.8 (13.4) | 3.5 (8.4)
  Systolic blood pressure: number analyzed (Participants) | 25 | 25
  Systolic blood pressure | 6.8 (11.9) | 5.8 (16.1)

64. Secondary Outcome: Change in Vital Signs (Pulse)
Description: Pulse was measured after a 5-minute rest in sitting position. Change from baseline (week 0) in pulse. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 208
Population: SAS. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
beats/min | -15.3 (14.2) | -3.8 (16.5)

65. Secondary Outcome: Change in Urinalysis (Protein, Glucose and Occult Blood)
Description: The urinalysis was the measurements of protein, glucose, and occult blood at baseline (within 4 weeks prior to week 0) and week 208 and categorised as negative, trace, 1+, 2+ and 3+. Number of participants in each category at baseline and week 208 are presented. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 208
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Participants
  Protein: Negative (Baseline) | 23 | 22
  Protein: Trace (Baseline) | 2 | 4
  Protein: 1+ (Baseline) | 0 | 0
  Protein: 2+ (Baseline) | 0 | 0
  Protein: 3+ (Baseline) | 0 | 0
  Protein: Negative (Week 208) | 17 | 18
  Protein: Trace (Week 208) | 8 | 7
  Protein: 1+ (Week 208) | 0 | 0
  Protein: 2+ (Week 208) | 0 | 1
  Protein: 3+ (Week 208) | 0 | 0
  Glucose: Negative (Baseline) | 25 | 26
  Glucose: Trace (Baseline) | 0 | 0
  Glucose: 1+ (Baseline) | 0 | 0
  Glucose: 2+ (Baseline) | 0 | 0
  Glucose: 3+ (Baseline) | 0 | 0
  Glucose: Negative (Week 208) | 25 | 26
  Glucose: Trace (Week 208) | 0 | 0
  Glucose: 1+ (Week 208) | 0 | 0
  Glucose: 2+ (Week 208) | 0 | 0
  Glucose: 3+ (Week 208) | 0 | 0
  Occult blood: Negative (Baseline) | 24 | 25
  Occult blood: Trace (Baseline) | 1 | 1
  Occult blood: 1+ (Baseline) | 0 | 0
  Occult blood: 2+ (Baseline) | 0 | 0
  Occult blood: 3+ (Baseline) | 0 | 0
  Occult blood: Negative (Week 208) | 24 | 22
  Occult blood: Trace (Week 208) | 1 | 2
  Occult blood: 1+ (Week 208) | 0 | 1
  Occult blood: 2+ (Week 208) | 0 | 0
  Occult blood: 3+ (Week 208) | 0 | 1

66. Secondary Outcome: Change in Blood Coagulation Test (Prothrombin Time and APTT)
Description: Change from baseline (within 4 weeks prior to week 0) in blood coagulation test parameters: prothrombin time and APTT. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 208
Population: SAS.
Measure: Median (Full Range); unit: sec
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
sec
  Prothrombin time | 0.70 [-0.3 to 2.4] | 1.20 [-0.2 to 2.2]
  APTT | 0.70 [-5.3 to 5.0] | 0.80 [-7.4 to 6.4]

67. Secondary Outcome: Change in ECG
Description: The ECG was recorded after a 3-minute rest in supine position at baseline (within 4 weeks prior to week 0) and week 208 and categorised as normal, abnormal NCS or abnormal CS. Number of participants in each ECG category at baseline and week 208 are presented. Missing values were imputed using the LOCF method.
Time Frame: Baseline, week 208
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | NN-220 0.033 mg/kg/Day | NN-220 0.066 mg/kg/Day
Number analyzed (Participants) | 25 | 26
Participants
  Normal (Baseline) | 15 | 14
  Abnormal NCS (Baseline) | 10 | 12
  Abnormal CS (Baseline) | 0 | 0
  Normal (Week 208) | 20 | 16
  Abnormal NCS (Week 208) | 5 | 9
  Abnormal CS (Week 208) | 0 | 1

ADVERSE EVENTS:
Time Frame: Week 0 to week 234 (208 weeks treatment period + 26 weeks extended treatment period) + 7 days (follow-up period).
Description: All presented AEs are TEAEs. A TEAE (for the entire trial) was defined as an event that had onset date on or after the date of visit 2 (week 0; start of treatment) and no later than 7 days after the last day of trial product administration. Results are based on the SAS, which included all participants receiving at least one dose of trial product.
Groups:
- 0.033 mg/kg/Day: Participants received s.c. injection of NN-220, 0.033 mg/kg/day once daily for 234 weeks (104 weeks of pivotal phase + 104 weeks of extension phase + 26 weeks extended treatment phase).
- 0.066 mg/kg/Day: Participants received s.c. injection of NN-220, 0.066 mg/kg/day once daily for 234 weeks (104 weeks of pivotal phase + 104 weeks of extension phase + 26 weeks extended treatment phase).
Arm/Group | 0.033 mg/kg/Day | 0.066 mg/kg/Day
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 9/25 | 10/26
Other Adverse Events (participants affected / at risk) | 24/25 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.033 mg/kg/Day (N=25) | 0.066 mg/kg/Day (N=26)
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Conductive deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Craniosynostosis (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Dental caries (Gastrointestinal disorders) | 2 (2) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Hamartoma (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Head banging (Psychiatric disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 1 (1)
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pulmonary artery therapeutic procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Supernumerary teeth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Testicular swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Velopharyngeal incompetence (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.033 mg/kg/Day (N=25) | 0.066 mg/kg/Day (N=26)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 3 (8)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (3)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 4 (5) | 7 (12)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 2 (2)
Chillblains (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Conjunctivitis (Infections and infestations) | 5 (6) | 6 (6)
Conjunctivitis allergic (Eye disorders) | 6 (11) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 3 (5)
Dental caries (Gastrointestinal disorders) | 4 (4) | 4 (11)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 7 (12) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 3 (4) | 8 (13)
Enteritis (Gastrointestinal disorders) | 2 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Gastroenteritis (Infections and infestations) | 8 (14) | 14 (33)
Gingivitis (Infections and infestations) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 6 (10) | 2 (5)
Hordeolum (Infections and infestations) | 1 (1) | 3 (5)
Hyperinsulinaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Impetigo (Infections and infestations) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 20 (34) | 18 (31)
Miliaria (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (10)
Molluscum contagiosum (Infections and infestations) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 19 (115) | 21 (121)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Otitis media (Infections and infestations) | 7 (9) | 8 (9)
Otitis media acute (Infections and infestations) | 4 (6) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (3) | 5 (6)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 9 (24) | 9 (12)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 4 (7)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Seasonal allergy (Immune system disorders) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 5 (14) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 5 (6)
Streptococcal infection (Infections and infestations) | 2 (3) | 3 (4)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 5 (9)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 8 (38) | 9 (43)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 7 (35) | 9 (30)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (8) | 2 (2)
Varicella (Infections and infestations) | 2 (2) | 5 (5)
Vomiting (Gastrointestinal disorders) | 4 (9) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT01927861/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-28): https://cdn.clinicaltrials.gov/large-docs/61/NCT01927861/SAP_001.pdf